CLINICAL TRIAL: NCT01232010
Title: Clinical Study to Investigate the Safety and Pharmacokinetics of Udenafil Tablet in Renal Impaired Male Patients
Brief Title: Clinical Study to Investigate the Safety and Pharmacokinetics of SK3530 Tablet in Renal Impaired Male Patients
Acronym: SK3530_RI_I
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: SK Chemicals Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Kyun-Seop Bae, Principal Investigator, Asan Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2007-0445
Record Dates: First submitted 2010-11-01; First posted 2010-11-02 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2015-01

CONDITIONS: Renal Insufficiency; Kidney Diseases; Urologic Diseases
Keywords: SK-3530; renal impairment; healthy volunteers
MeSH Terms: conditions — Renal Insufficiency; Kidney Diseases; Urologic Diseases | interventions — mirodenafil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy Volunteers (Experimental)
  Interventions: Drug: Mirodenafil
- Patients with severe renal impairment (Experimental)
  Interventions: Drug: Mirodenafil

INTERVENTIONS:
Drug: Mirodenafil — 50mg Single Oral Dose of

SUMMARY:
This study is designed to investigate the effect of renal impairment on the safety and pharmacokinetics of SK3530 in subjects with renal impairment compared to healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Adult males aged 19 to 64 years at screening.
* Subjects with body weight ≥ 50 kg and within ±30% of the ideal body weight : Ideal body weight = (height [cm] - 100)x0.9.
* Subjects who have received and understood completely the information regarding the current study and given written informed consents to voluntarily participate in the study and followed all instructions specified in the protocol.

Exclusion Criteria:

* Subjects with the test results of QTc > 430 ms or non-sinus cardiac rhythm by ECG analysis.
* Subjects with hypotension or hypertension.
* Subjects deemed ineligible by investigator based on other reasons, including abnormal laboratory values or diseases.

Ages: 19 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2009-11; Primary Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (AUC and Cmax) | 2days

CONTACTS AND LOCATIONS:
Overall Officials: Kyun-Seop Bae, M.D., Ph.D., Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- See also: Clinical Research Center, Asan Medical Center — http://crc.amc.seoul.kr